CLINICAL TRIAL: NCT05709314
Title: A Phase 2, Open-Label Study of AMDX-2011P as a Retinal Tracer in Participants With Cerebral Amyloid Angiopathy (CAA)
Brief Title: A Study of AMDX-2011P in Participants With CAA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amydis Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMDX-2011P-001; 5SB1AG073029-02 (NIH)
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Amyloid Angiopathy
Keywords: CAA
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Intervention Model Description: Phase 2, open-label, single arm, masked endpoint multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMDX-2011P 100 mg (Experimental): AMDX2011P 100mg (4ml) single bolus injection intravenous for diagnostic review
  Interventions: Drug: AMDX-2011P

INTERVENTIONS:
Drug: AMDX-2011P — AMDX-2011P single bolus injection intravenous for diagnostic review

SUMMARY:
The purpose of this study is to assess safety, tolerability, plasma pharmacokinetics and biologic activity of a single intravenous dose of AMDX-2011P in participants with cerebral amyloid angiopathy (CAA).

DETAILED DESCRIPTION:
This open-label, masked endpoint assessment study will evaluate the safety, tolerability, plasma pharmacokinetics (PK) and biological activity of an intravenous (IV) dose of AMDX-2011P in participants with CAA. Assessments of retinal images will be conducted by central masked assessors.

Participants will be admitted to the study site where eye examination and retinal imaging will be conducted before administration of the study drug. AMDX-2011P will be administered through a single IV bolus injection followed by safety assessments, retinal imaging and PK blood collection.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hereditary CAA or probable and definite symptomatic or asymptomatic sporadic CAA diagnosed through genetic testing or according to the modified Boston neuroradiological criteria, who had undergone at least one brain magnetic resonance imaging (MRI)prior to entry into study.
2. Abnormality consistent with CAA on historical MRI.
3. In general good health

Exclusion Criteria:

1. Presence of any underlying physical or psychological medical condition that, in the opinion of the investigator, would make it unlikely that the participant will complete the study per protocol.
2. Clinically significant laboratory abnormalities assessed by the investigator.
3. Active malignancy and/or history of malignancy in the past 5 years, with the exception of completely excised non-melanoma skin cancer or low-grade cervical intraepithelial neoplasia.
4. Prolonged QTcF (>450 ms for males and >470 ms for females),cardiac arrhythmia, or any clinically significant abnormality in the resting ECG, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
AMDX-2011P Adverse Events Profile | 8 days
  Incidence, nature and severity of AEs/SAEs

SECONDARY OUTCOMES:
Concentration of AMDX-2011P | 2 hours
  Plasma PK Concentration (CMax)AMDX-2011P to AMDX-2011
Pharmacokinetic Analysis of AMDX-2011P | 2 hours
  Area under the plasma versus time curve (AUC)
Biological Activity | 8 days
  Detection of amyloid deposits in the retina after intravenous AMDX-2011P administration using a conventional retinal fundus fluorescence imaging device.

CONTACTS AND LOCATIONS:
Overall Officials: David Bingaman, DVM, PhD, Study Director — Amydis Inc.
Locations (3):
- United States (3):
  - Associated Retina Consultants, Phoenix, Arizona
  - Global Research Management, Glendale, California
  - Eye Research Foundation, Newport Beach, California

IPD SHARING:
Plan to Share IPD: No